CLINICAL TRIAL: NCT04232891
Title: Early Detection of Relapses in Stage IV Colorectal Cancer Patients: REDCLOUD (REsidual Disease, Colorectal Cancer, Liquid biOpsy Detection)
Brief Title: Early Detection of Relapses in Stage IV Colorectal Cancer Patients
Acronym: REDCLOUD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fondazione del Piemonte per l'Oncologia (Other)
Responsible Party: Sponsor
Other Study IDs: 017-FPO18
Record Dates: First submitted 2020-01-14; First posted 2020-01-18 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Metastatic Colorectal Cancer
Keywords: liquid biopsy; metastatic colorectal cancer; early detection of metastases
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Liquid Biopsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: liquid biopsy — detection of tumor DNA alteration in cf-DNA

SUMMARY:
This study is a prospective, multicenter, observational study on metastatic, operable colorectal cancer to evaluate the proof of concept of the cfDNA analysis for the early detection of recurrences

ELIGIBILITY:
Inclusion Criteria:

1. Histological confirmed adenocarcinoma of the colon or rectum with synchronous metastatic disease (localized in liver or in liver and lung) eligible for surgery immediately or after neo-adjuvant treatment.
2. Planned primary treatment at one of the REDCLOUD participating hospital centers.
3. Evidence of at least one measurable lesion, as per RECIST 1.1.
4. Male or female ≥ 18 years of age at time of informed consent.
5. Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1. No prior chemotherapy neither for localized nor for metastatic disease.
6. No major comorbidities that would preclude the compliance with the planned therapeutic program as judged by the Investigator.
7. Life expectancy > 3 months.
8. Availability of biological samples (blood and tumor tissue).
9. Patients enrolled in local prospective protocols, in which samples have been collected according REDCLOUD procedures may be included.
10. Signed and dated informed consent.

Exclusion Criteria:

1. Any physical or medical condition that would contraindicate chemotherapy and/or surgery.
2. Any other metastatic site, except for liver and lung metastases
3. Transplant recipients
4. Known history of human immunodeficiency virus (HIV) infection. Note: HIV testing will only be conducted in jurisdictions specifically requiring it.
5. Known active hepatitis B or hepatitis C infection.
6. Pregnant or lactating women
7. Other co-existing malignancies or malignancies diagnosed within the last 5 years with the exception of localized basal and squamous cell carcinoma or cervical cancer in situ adequately treated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Metastatic colorectal cancer patients eligible to metastasectomy
Sampling Method: Non-Probability Sample
Enrollment: 141 (Estimated)
Dates: Start 2019-11-18 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
relapse rate in MRD+ patients | immediately surgery and up to 2 years after surgery
  Percentage of patients with MRD (minimal residual disease) with documented relapse. MRD is defined as detection, through liquid biopsy, of any of the molecular alterations evaluated in any plasma sample drawn within 40 days from surgery.
relapse rate in MRD- patients | immediately surgery and up to 2 years after surgery
  Percentage of patients with no MRD (minimal residual disease) with documented relapse. MRD- is defined as detection, through liquid biopsy, of no molecular alterations evaluated in any plasma sample drawn within 40 days from surgery.

SECONDARY OUTCOMES:
minimal residual disease detection rate | up to 40 days after surgery
  percentage of patients with detectable MRD (minimal residual disease) defined as detection, through liquid biopsy, of any of the molecular alterations evaluated in any plasma sample drawn within 40 days from surgery.

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Fondazione del Piemonte per l' Oncologia - IRCCS Candiolo, Candiolo, Torino
  - Ospedale Mauriziano, Torino

IPD SHARING:
Plan to Share IPD: Undecided